CLINICAL TRIAL: NCT02489110
Title: Webnovela for Hispanic Dementia Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Stanford University (Other)
Responsible Party: Principal Investigator, Bruno Kajiyama, CEO, Photozig, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pz-A104a; R44AG041552 (NIH)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's Disease; Dementia; caregiving; caregiver; coping; coping with caregiving; stress; Hispanic caregiver; Latino caregiver
MeSH Terms: conditions — Alzheimer Disease; Dementia

ARMS (2):
- Webnovela (Experimental): Caregivers will watch the Webnovela and read related information. The Webnovela is a short online Telenovela in Spanish, specifically designed for Hispanic caregivers on how to cope with dementia caregiving. A DVD will be available to participants without Internet access.
  Interventions: Behavioral: Webnovela
- Control (Active Comparator): Caregivers will be directed to existing web sites, such as NIA Alzheimer's and Dementia Resources in Spanish. Participants will receive related materials in Spanish language.
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Webnovela
  Arms: Webnovela
Behavioral: Information
  Arms: Control

SUMMARY:
Photozig and Stanford University are creating a new program for Hispanic dementia caregivers to help cope with caregiving, alleviate related stress, and enhance quality of life for caregivers, with funding from the National Institute on Aging. The program includes a new education online telenovela (Webnovela), online resources, handouts and a DVD (for users without Internet) on how to deal with caregiving stress and handle difficult situations.

DETAILED DESCRIPTION:
The goal of Webnovela program is to evaluate and develop materials for helping caregivers to cope with caregiving, alleviate related distress, and improve their quality of life.

The investigators are evaluating different materials, which may provide caregiving strategies, practical tips and help to enhance caregivers' skills to deal with demanding tasks of caregiving, alleviate related stress, and improve quality of life.

Research Program Steps:

1. Caregivers will be asked some simple questions about themselves and their family members to see if they are eligible for the project (fill out Enrollment Form and Informed Consent).
2. A Program survey will be sent, which can be completed online, or returned in a pre-mailed envelope.
3. Participants will receive links to online resources, related materials and instructions. The investigators ask participants to access the online resources, read provided brochures and guides, and follow the instructions. Materials are expected to help participants in their caregiver role.
4. After completing the program, the second and final survey should be filled out online or returned by pre-mailed envelope.

ELIGIBILITY:
Inclusion Criteria:

* Care for an individual with Alzheimer's Disease or other dementia.
* Have Internet access or own a DVD player.
* Minimum age of 18 years old.
* Belong to Hispanic/Latino ethnic group.
* Spend at least 8 hours/week caring for a person with dementia, which may include assisting, watching, monitoring, or being available to help (e.g. during sleep time)

Exclusion Criteria:

* Severe psychological or physical illness.
* Inability to read and follow Spanish instructions.
* High level of depressive symptoms.
* Unwillingness to participate in all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Kajiyama, MS, Principal Investigator — Photozig, Inc.
Locations (1):
- Photozig, Inc., Moffett Field, California, United States

REFERENCES:
- See also: Dementia Caregiving Program for Hispanic caregivers — http://www.miramirela.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Webnovela: Caregivers will watch the Webnovela and read related information. The Webnovela is a short online Telenovela in Spanish, specifically designed for Hispanic caregivers on how to cope with dementia caregiving. A DVD will be available to participants without Internet access.
  Webnovela
- Control: Caregivers will be directed to existing web sites, such as NIA Alzheimer's and Dementia Resources in Spanish. Participants will receive related materials in Spanish language.
  Information
Period: Overall Study
Arm/Group | Webnovela | Control
Started | 75 | 75
Completed | 48 | 50
Not Completed | 27 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Webnovela | Control | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.2) | 51.5 (9.4) | 52.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 129
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 75 | 150
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stress on the Perceived Stress Scale
Description: The "Perceived Stress Scale" measures the overall level of stress. This instrument contains 10 items accessing overall appraisals of stress in the past month. Minimum score (best value)=0. Maximum score (worst value)=40. Higher values represent a worse outcome.
Time Frame: 3 months
Population: One (1) subject in the Webnovela group and one (1) subject in the Control group completed the study, but they did not have full data related to the Primary Outcome "Stress on the Perceived Stress Scale." These subjects were not included in this data analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Webnovela | Control
Number analyzed (Participants) | 47 | 49
units on a scale | 14.57 (5.54) | 15.37 (5.89)

2. Secondary Outcome: Caregiver Burden on the Revised Memory and Behavior Problems Checklist
Description: This scale measures the type/number of dementia patients disturbing behaviors, and how much they bother caregivers with 24 items describing possible troublesome behaviors that the patient might evidence in the past month. Caregivers are first asked whether the dementia patient had displayed any of these in the time period, and secondly to rate on a 5-point scale (0=not at all; 4= extremely) how much this "bothered or upset" them. A "conditional bother" score is calculated which is the "upset" or "bother" ratings for only the problematic behavior that occurred. The scale refers to the caregiver. Minimum score (best value)=0. Maximum score (worst value)=4. Higher values represent a worse outcome.
Time Frame: 3 months
Population: Two (2) subjects in the Webnovela group completed the study, but they did not have full data related to the Secondary Outcome "Caregiver Burden on the Revised Memory and Behavior Problems Checklist." These subjects were not included in this data analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Webnovela | Control
Number analyzed (Participants) | 46 | 50
units on a scale | 0.51 (0.57) | 0.60 (0.86)

ADVERSE EVENTS:
Arm/Group | Webnovela | Control
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes